CLINICAL TRIAL: NCT06665659
Title: Retrospective Evaluation of the Tecnis Eyhance and OphthalmoPro Zoe Intraocular Lenses
Brief Title: Evaluation of the Eyhance and Zoe Lenses
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: Southend NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 345720
Record Dates: First submitted 2024-08-15; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Monofocal IOL group: Participants who have had either the Tecnis Eyhance or OphthalmoPro Zoe monofocal lens implanted during routine cataract surgery

SUMMARY:
The goal of this observational study is to assess distance and near visual acuity of patients who have undergone cataract surgery with two intraocular lenses (IOLs). The main outcomes are:

To assess distance and near visual acuity of patients who have undergone cataract surgery with two intraocular lenses (IOLs) To assess depth of focus of the IOLs To assess tilt and decentration of the IOLs

The potential participants will be chosen from the list of patients in the Southend NHS database who have had routine cataract surgery using the Zoe or Eyhance lenses in the past 12 months and contacted by phone and letter. The member of the ophthalmological team carrying out the screening will use the research inclusion and exclusion criteria to identify 50 potential participants. Once identified, the potential participants will be asked if they would be willing to discuss inclusion into the study with a member of the clinical care team (Prof Myerscough or Dr Law). If they agree, they will be asked to attend one further clinical visit.

They will be given a patient information sheet and consent form at this visit. All potential participants will be informed that participation in this research study will be entirely voluntary.

At the clinical visit participants will have their vision assessed, have dilating drops instilled, and undergo two non-invasive scans of their eyes.

DETAILED DESCRIPTION:
Background and rationale:

Artificial lenses, otherwise known as intraocular lenses (IOLs), are used to replace the natural crystalline lens within the eye during cataract or refractive lens surgery. Monofocal IOLs are the traditional IOL type and provide excellent distance vision following cataract surgery, however spectacles are required for reading and intermediate distance tasks.

The evolution of IOLs has been rapid over the last 50 years and there are now monofocal IOLs on the market (available to NHS hospitals) which aim to improve intermediate (computer distance) vision by increasing depth of focus.

There is currently little evidence to support which optical design provides the best visual outcome and existing literature for visual outcomes of intraocular lenses are largely derived from either ex-vivo bench studies, or tightly controlled groups in research settings with far reaching exclusion criteria. The idea of this retrospective study was to provide more data on how lenses perform in a busy NHS corneal service, not excluding (most) corneal comorbidity. The study aims to evaluate two of the monofocal IOLs that have been routinely used at Southend NHS hospital.

This research project is a retrospective study involving 50 subjects who have already received one of two standard treatment monofocal IOLs; the Ophthalmo Pro Zoe and the Tecnis Eyhance. Potential participants will be invited to attend an additional study visit at the hospital where their visual outcomes will be evaluated. There will be no comparison between the lenses therefore there is no need to match the participants or split the groups evenly.

Patient recruitment:

Both the Tecnis Eyhance and OphthalmoPro Zoe are monofocal lenses approved for use in patients having routine cataract surgery and are available in the Southend Eye Clinic lens bank. Of these patients 50 participants who have had routine cataract surgery with one of these lenses within the past 12 months will be chosen. Patients will be identified from the Southend NHS database. The database search will be carried out by the clinical care team. Potential participants will be asked to come to the eye clinic for one additional follow up visit in which they will have vision assessed in the operated eye(s). Potential participants will be contacted by phone and by letter.

Each participant will be expected to be part of the study for the duration of one hospital visit. This post-surgical assessment will be within 18 months after surgery. This will mark the end of their participation required. The visit should last up to 45 minutes.

Informed consent for study involvement will be secured at the follow up visit for those who agree to participate. Three copies of the consent form will be filled out. One copy will be retained by the patient (with a copy of the patient information sheet), the other by the investigators and the last will be kept in the patient's NHS file. At the point of consent during the follow up visit the subject will be assigned a subject number code.

Participants will be free to withdraw from the study at any time but any data already collected will be included.

Risk, burden and benefit to participants:

The study will include one additional visit. As a result, participation in this study will increase the length and number of appointments that the participant will have to attend. The additional appointment will allow additional care and screening for the participant.

Assessment will involve dilation of the pupils by eye drops. This occurs as part of the routine pre- and post-surgical assessments normally. The co-investigators (Prof Myerscough and Dr Law) carrying out this assessment are an ophthalmic surgeon and a registered Optometrist respectively and dilation and the use of mydriatics is a routine procedure.

All assessments carried out in this study are noncontact and non-invasive. Scans of the eye do not use any radiation. Participants may experience some light sensitivity during the examination, but this is the same as they would have experienced at previous appointments and does not cause any lasting damage.

There is a minimal risk of raised intraocular pressure following the application of dilating drops. However, the participants would have already had this done as a part of their pre-operative visit without any side effects. The risk of this side effect is minimised further by removal of the cataract therefore the risk of raised intraocular pressure at the postoperative visit is negligible.

The participants will benefit from an additional follow up visit, as this will increase the monitoring and care for any post-surgical complications compared to usual practice. They will have the opportunity to ask questions to the optometrist and ophthalmologist about their eye condition. It will also help increase the patient awareness and understanding of the surgical procedure and outcomes.

Ethical approval:

The protocol, informed consent form, participant information sheet and any proposed advertising material will be submitted to an appropriate Research Ethics Committee (REC), and host institution for written approval. The Investigator will submit and, where necessary, obtain approval from the above parties for all substantial amendments to the original approved documents.

Funding:

There is no external funding application.

Publication policy and data management:

No identifiable personal data will be used in any publications. If participants have expressed an interest in the results of the study, they will be sent a lay summary of the results and outcomes.

The scientific quality of the research will be assessed within the co-investigator's institution and the educational supervisor. The study forms part of an MD project and hence has been subject to review by the education supervisors, the research team and the university ethics council. The statistics will be reviewed by the educational supervisor.

The results of the study will be disseminated in peer reviewed scientific journals, internal reports, and at conference presentations.

As with all studies, there is a very small risk of breach in confidentiality and failure to maintain data securely. However, every care will be taken to ensure that a strict policy of data protection and securing of the data is followed by any members of the study who are all qualified clinicians and familiar with this policy.

The co-investigators (Prof Myerscough and Dr Law) are part of the Ophthalmological clinical care team. These team members have access to the data as part of the clinical record keeping required for routine NHS assessment and care. There is no referral to an outside research team and no other investigators will have access to any personal data. If the patient agrees to participate then they will be made fully aware that their details will be reviewed and are free to decline, in which case their records will not be included in the process.

To maintain anonymity, participant data will be identified only by a code, which will be entered on to a password protected spreadsheet on the NHS database and will only be accessible to the coinvestigators, Prof Myerscough and Dr Law, both of whom are part of the Southend Ophthalmological clinical care team and are bound by a code of conduct and data protection. No personal data will be removed or transcribed from the patient records. Initial examination findings from the postoperative visit will be entered into written patient notes, which will be later scanned and uploaded on to the NHS database and then destroyed, as is protocol for all patient notes in the ophthalmology department at Southend Hospital. All data will be stored using OneDrive. No data will be stored on the desktop or on any external hard drives that may be accessed by anyone else.

Plymouth University is the Sponsor and will be the data controller for the study. The Mid and South Essex NHS trust (to which Southend Hospital belongs), the sponsor representative from Plymouth University, and regulatory bodies will have access to data to ensure that the study is being run correctly. Dr Sharma will be analysing the anonymised data at Plymouth University and will not have access to patient identifiable information or patient notes. Any data that leaves Southend Hospital will be anonymised before being shared with the research team via OneDrive.

Informed consent will be obtained from each individual participant. A signed copy of the consent form will be kept by the subject, the investigators and one will be kept in the patient file. They are all required to be consenting adults with mental capacity, who can show that they are able to understand the patient information sheet and consent to the study themselves. It will be collected on by one of the two investigators (Prof Myerscough or Dr Law) at the follow up visit post procedure.

If the participant is unable to communicate adequately to the investigators, then they will be classified as unable to give valid informed consent to the study.

The participant will be withdrawn from the study if it is felt that they no longer has the capacity to give informed consent for the study. They will need to be compliant with the assessment and follow up appointment to complete the study. If they are withdrawn it will not affect their surgery or medical care by the hospital. All the data gathered prior to the withdrawal will be removed from the study and destroyed. This is unlikely to happen as participants will only need to attend for one visit, after which there would be no further contact with them. Participants who cannot give consent to attend this visit will not be included.

The data will be archived at Plymouth University for 10 years.

Postoperative visit routine:

At the visit the following non-invasive visual function tests will be conducted:

* A detailed assessment of visual acuity
* An objective and subjective assessment of refraction will be used to determine if there is any residual refractive error.
* Defocus curve profiles (visual acuity over imposed defocus) will be measured for each patient over a defocus range of +1.50D to -4.00D in 0.50D steps. The presentation of the letters and lenses will be randomised.

The MS-39 (CSO Ophthalmic) will be used to determine the position of the IOL and to assess if any tilt or decentration is present.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18) patients with cataract requiring cataract surgery with phacoemulsification and intraocular lens implantation.
* Patients who have had either an OphthalmoPro Zoe or a Tecnis Eyhance monofocal lens implanted during routine cataract surgery within the past year

Exclusion Criteria:

* Previous penetrating keratoplasty or anterior lamellar keratoplasty
* Patients who are not willing to cooperate for the follow up period
* Patients where it is not possible to take informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both the Tecnis Eyhance and OphthalmoPro Zoe are monofocal lenses approved for use in patients having routine cataract surgery and are available in the Southend Eye Clinic lens bank. Of these patients 50 participants who have had routine cataract surgery with one of these lenses within the past 12 months will be chosen. Patients will be identified from the Southend NHS database. The database search will be carried out by the clinical care team. Potential participants will be asked to come to the eye clinic for one additional follow up visit in which they will have vision assessed in the operated eye(s). Potential participants will be contacted by phone and by letter.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | From enrollment to the clinical assessment at 3 months
  To assess distance and near visual acuity of patients who have undergone cataract surgery with two intraocular lenses (IOLs)

SECONDARY OUTCOMES:
Depth of focus | From enrollment to the clinical assessment at 3 months
  To assess depth of focus of the IOLs
Tilt | From enrollment to the clinical assessment at 3 months
  To assess tilt of the IOLs
Decentration | From enrollment to the postoperative visit at 3 months
  To assess decentration of the IOLs

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Buckhurst, PhD, Study Director — Plymouth University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lapp T, Wacker K, Heinz C, Maier P, Eberwein P, Reinhard T. Cataract Surgery-Indications, Techniques, and Intraocular Lens Selection. Dtsch Arztebl Int. 2023 May 30;120(21):377-386. doi: 10.3238/arztebl.m2023.0028. PMID 36794457
- [Background] Kanclerz P, Toto F, Grzybowski A, Alio JL. Extended Depth-of-Field Intraocular Lenses: An Update. Asia Pac J Ophthalmol (Phila). 2020 May-Jun;9(3):194-202. doi: 10.1097/APO.0000000000000296. PMID 32511121